CLINICAL TRIAL: NCT02695472
Title: A Phase 2, Double-Blind, Placebo-Controlled Study of NSI-189, a Neurogenic Compound Among Out-Patients With Major Depressive Disorder
Brief Title: Study of NSI-189 for Major Depressive Disorder
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Neuralstem Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NS2014-1
Record Dates: First submitted 2016-02-15; First posted 2016-03-01 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-02

CONDITIONS: Major Depressive Disorder
Keywords: Depression; Major Depressive Disorder (MDD); Major Depressive Disorder; Neurogenesis; Synaptogenesis; NSI-189; Neuralstem
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — BID protein, human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Placebo Arm (Placebo Comparator): One Placebo tablet, twice daily
  Interventions: Drug: Placebo
- 40 Milligrams NSI-189, total dose daily (Experimental): One 40 Milligrams NSI-189 tablet and 1 placebo tablet per day
  Interventions: Drug: Placebo; Drug: 40 Milligrams NSI-189
- 80 Milligrams NSI-189, total dose daily (Experimental): One 40 Milligrams NSI-189 tablet twice per day
  Interventions: Drug: 80 Milligrams NSI-189

INTERVENTIONS:
Drug: 80 Milligrams NSI-189 — Orally Administered
  Other Names: NSI-189 twice per day (BID)
  Arms: 80 Milligrams NSI-189, total dose daily
Drug: Placebo — Orally administered
  Arms: 40 Milligrams NSI-189, total dose daily; Placebo Arm
Drug: 40 Milligrams NSI-189 — Orally Administered
  Other Names: NSI-189 Once a day (QD)
  Arms: 40 Milligrams NSI-189, total dose daily

SUMMARY:
The study will consist of a screening period and a randomized treatment. Approximately 220 subjects who meet eligibility during the screening period will be randomized to initiate a 12-week, double-blind treatment with NSI-189 80 milligrams/day (provided as 40 milligrams twice per day), NSI-189 40 milligrams once a day, or placebo.

DETAILED DESCRIPTION:
The screening period will range from a minimum of 14 days to a maximum of 28 days. The Investigators will determine that the subjects meet eligibility criteria and will collect the demographic and medical data permitting full characterization of the subject.

The duration of the randomization period will be 12 weeks. Subjects who meet inclusion/exclusion criteria at the Baseline Visit will be randomized to NSI-189 80 milligrams/day, given as 40 milligrams twice per day, NSI-189 40 milligrams/day, given once a day, or placebo. The treatment will be double-blinded.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has the ability to understand the purpose, potential benefits and risks of the study and to provide signed and dated informed consent, authorizing the use of protected health information in accordance with national and local Subject privacy regulations.
2. Males and females 18 to 60 years of age, inclusive, at the time of informed consent.
3. Diagnosis of major depressive disorder, recurrent, as per Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria and confirmed by Structured Clinical Interview for the Diagnostic and Statistical Manual specific for Clinical Trials. Their major depressive episode must be at least 8 weeks in duration and confirmed via Structured Clinical Interview for the Diagnostic and Statistical Manual mood module interview administered by a remote, independent raters, prior to the baseline visit.
4. Montgomery-Asberg Depression Scale (MADRS) score of 20 or greater, at Screening and Baseline (MADRS score confirmed to be 20 or greater via remote SAFER interview by an independent rater prior to the baseline visit).
5. The following applies to female Subjects: Non-pregnant, non-lactating females of childbearing potential are eligible as long as they agree to use a double barrier method of birth control from Screening until 3 months following discontinuation of IP. Women who are not of childbearing potential (bilateral oophorectomy, bilateral tubal ligation, hysterectomy, or post-menopausal for at least 1 year) will not require such parameters in order to be eligible.
6. The following applies to male subjects: Male subjects with a female partner of childbearing potential will be required to use double barrier method of birth control or practice abstinence during this study and for 3 months following discontinuation of Investigational Product. Note: These requirements also apply for male subjects who have had a vasectomy.
7. Body mass index (BMI) ≥19.5 and ≤38.0 kg/m2, at Screening. Bodyweight must be >50 kg.
8. Of stable medical health, in the opinion of the Site Investigator, as determined by Investigator discretion (medical history, physical examination, vital signs, ECG, and clinical laboratory assessments).

Exclusion Criteria:

1. Clinically significant history or evidence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, neurological, immunological, or other major disease as determined by the Investigator or designee such that participation in the study would place subjects at increased risk for serious adverse events.
2. History of cancer or malignancy within the last 5 years. Note: Subjects with basal or squamous cell carcinoma may be permitted into the study on a case by case basis.
3. History of seizures; head trauma; or any clinically significant finding on the neurologic examination such that participation in the study would place subjects at increased risk for serious adverse events.
4. Previous or current diagnosis of bipolar or schizoaffective disorder or psychotic disorder, or any psychotic symptoms during the current major depressive episode (according to Diagnostic and Statistical Manual of Mental Disorders, 5th edition).
5. Subjects who have a concurrent primary psychiatric diagnosis, diagnosed by Structured Clinical Interview for Diagnostic and Statistical Manual of Mental Disorders, 5th edition, other than depression.
6. Subjects with delirium, dementia, Parkinson's disease, or Huntington's disease.
7. Subjects who have failed to respond to more than two antidepressant trials of adequate dose (as defined in Massachusetts General Hospital Antidepressant Treatment Response) and duration (at least 8 weeks in duration) during the current major depressive episode as determined by the local rater and confirmed by an independent, remote rater prior to the baseline visit.
8. Subjects with clinically significant suicidal ideation and/or behavior currently as determined by the Site Investigator, such that participation in the study would place subjects at increased risk for serious adverse events.
9. Subjects with any current homicidal ideation.
10. Clinically significant abnormal clinical chemistry values, as determined by the Site Investigator, or any values for Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), total bilirubin or creatinine that are 1.5 times above the upper limit of normal (ULN) and deemed clinically significant by the Site Investigator; any clinically significant values as determined by the Site Investigator for platelets or hemoglobin that are below the lower limit of normal (LLN); or any out of normal range values for white blood cells (WBC) deemed clinically significant by the Site Investigator.
11. Clinically significant (as determined by the Investigator) 12-lead Electrocardiogram (ECG) abnormalities, including corrected QT interval using Bazett's correction method of >450 msec for males and >470 msec for females.
12. Subjects with (current) severe Post-Traumatic Stress Disorder (PTSD), severe Obsessive Compulsive Disorder (OCD), severe binge eating disorder, or subjects with anorexia or bulimia nervosa active within the past three years.
13. Subjects who plan to undergo elective invasive procedures/surgeries at any time during the study through End-of-study.
14. Subjects taking excluded medications (See Appendix 1)..
15. History of alcohol or drug-dependence or abuse by Diagnostic and Statistical Manual of Mental Disorders, 5th edition criteria and confirmed by Structured Clinical Interview for the Diagnostic and Statistical Manual specific for Clinical Trials within 12 months prior to Screening.
16. Positive screening test or baseline test for drugs-of-abuse (cocaine, amphetamines, barbiturates, opiates, benzodiazepines, cannabinoids, phencyclidine). Note any positive test result(s) for benzodiazepine(s), opiates, or psychostimulants accompanied by confirmation of a prescription for a valid medical reason will be allowed.
17. Positive serum β-human chorionic gonadotropin (β-HCG) test at Screening or positive urine pregnancy test at baseline that is consistent with pregnancy (females only).
18. Donation or loss of whole blood >200 mL within 30 days prior to dosing or ≥500 mL within 56 days prior to dosing. Note: Blood taken for routine medical evaluations totaling less than 50 mL will be permitted.
19. Females who are pregnant, lactating, or planning to become pregnant during the study.
20. Does not tolerate venipuncture.
21. Subjects who have had electroconvulsive therapy within the 6 months prior to Screening.
22. Current enrollment in any other drug, biologic, device, or clinical study, or treatment with an Investigational Product or approved therapy for investigational use within 45 days (or 5 half-lives, whichever is longer) prior to Day 1 of Investigational Product administration.
23. Any concurrent disease or condition that, in the opinion of the Investigator, would make the subject unsuitable for participation in the clinical study.
24. Subject who, in the opinion of the Site Investigator, are unable to understand the protocol requirements, instructions and study-related restrictions, the nature, scope and possible consequences of the clinical study.
25. Subject who, in the opinion of the Site Investigator, are unlikely to comply with the protocol requirements, instructions and study-related restrictions; e.g., uncooperative attitude, inability to return for follow-up and improbability of completing the clinical study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 220 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Montgomery-Asberg Depression Rating Scale (MADRS) | Up to 12 weeks

SECONDARY OUTCOMES:
Symptoms of Depression Questionnaire (SDQ) | Up to 12 weeks
The Massachusetts General Hospital Cognitive and Physical Functioning Questionnaire (MGH CPFQ) | Up to 12 weeks
17-item Hamilton Rating Scale for Depression (HAMD17) | Up to 12 weeks
Clinical Global Impressions - Severity and Improvement (CGI-S, CGI-I) | Up to 12 weeks
Cogstate Brief Battery | Up to 12 weeks
  A computerized battery used to measure psychomotor, attention, learning and working memory performance. The subject results are compared with normative data from a population with similar age and gender.
CogScreen | Up to 12 weeks
  A computerized battery focused on measures of attention, concentration, information processing, memory span, and working memory. The subject results are compared with normative data from a population with similar age and gender.

CONTACTS AND LOCATIONS:
Overall Officials: Karl Johe, Ph.D., Study Director — Neuralstem Inc.
Locations (13):
- United States (13):
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - Synergy San Diego, National City, California
  - Clinical Trials of the Rockies, Denver, Colorado
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Clinical Neuroscience Solutions, Inc, Orlando, Florida
  - Institute for Advanced Medical Research, Alpharetta, Georgia
  - Psychiatric Medicine Associates, LLC, Skokie, Illinois
  - St. Louis Clinical Trials, LC, St Louis, Missouri
  - Richmond Behavioral Associates, Staten Island, New York
  - Midwest Clinical Research Center, LLC, Dayton, Ohio
  - Clinical Neuroscience Solutions, Inc., Memphis, Tennessee
  - FutureSearch Trials of Dallas, Dallas, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Fava M, Johe K, Ereshefsky L, Gertsik LG, English BA, Bilello JA, Thurmond LM, Johnstone J, Dickerson BC, Makris N, Hoeppner BB, Flynn M, Mischoulon D, Kinrys G, Freeman MP. A Phase 1B, randomized, double blind, placebo controlled, multiple-dose escalation study of NSI-189 phosphate, a neurogenic compound, in depressed patients. Mol Psychiatry. 2016 Oct;21(10):1372-80. doi: 10.1038/mp.2015.178. Epub 2015 Dec 8. PMID 26643541
- [Derived] Tajiri N, Quach DM, Kaneko Y, Wu S, Lee D, Lam T, Hayama KL, Hazel TG, Johe K, Wu MC, Borlongan CV. NSI-189, a small molecule with neurogenic properties, exerts behavioral, and neurostructural benefits in stroke rats. J Cell Physiol. 2017 Oct;232(10):2731-2740. doi: 10.1002/jcp.25847. Epub 2017 Apr 25. PMID 28181668